CLINICAL TRIAL: NCT06880016
Title: Evaluation of Serial Lung Ultrasound Data After Surfactant Treatments Applied With Different Methods in Preterm Babies
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Konya City Hospital (Other)
Responsible Party: Principal Investigator, Melek Buyukeren, Associate Professor, Konya City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: KSH_MB_2025_3
Record Dates: First submitted 2025-03-11; First posted 2025-03-17 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-03

CONDITIONS: Newborn Complication; Respiratory Distress Syndrome, Newborn
Keywords: NEWBORN; Respiratory Distress Syndrome; surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Distress Syndrome

STUDY DESIGN:
Intervention Model Description: The first method involves intubating the infant, administering intratracheal surfactant, and then extubating them back to nasal respiratory support (ENSURE method). The second method involves delivering surfactant via a thin catheter (5F) directly into the trachea while the infant remains on existing nasal respiratory support, without disconnecting them from it (LISA method).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ensure group (Experimental): The first method involves intubating the infant, administering intratracheal surfactant, and then extubating them back to nasal respiratory support (ENSURE method).
  Interventions: Diagnostic Test: Evaluation of serial lung ultrasound data after ENSURE surfactant treatments
- Lisa group (Experimental): The second method involves delivering surfactant via a thin catheter (5F) directly into the trachea while the infant remains on existing nasal respiratory support, without disconnecting them from it (LISA method).
  Interventions: Diagnostic Test: Evaluation of serial lung ultrasound data after LISA surfactant treatments

INTERVENTIONS:
Diagnostic Test: Evaluation of serial lung ultrasound data after ENSURE surfactant treatments — Intubating the infant, administering intratracheal surfactant, and then extubating them back to nasal respiratory support (ENSURE method)
  Arms: Ensure group
Diagnostic Test: Evaluation of serial lung ultrasound data after LISA surfactant treatments — Delivering surfactant via a thin catheter (5F) directly into the trachea while the infant remains on existing nasal respiratory support, without disconnecting them from it (LISA method)
  Arms: Lisa group

SUMMARY:
This study aims to investigate the relationship between the method of surfactant administration and improvements in serial lung ultrasound findings in preterm infants requiring surfactant therapy.

DETAILED DESCRIPTION:
In the neonatal intensive care unit, lung ultrasound was first used for the diagnosis of neonatal respiratory distress syndrome (RDS) by Avni et al. in 1990. Following this, lung ultrasound rapidly became widespread in neonatal intensive care units and was seen as a potential alternative to chest X-rays. It is now frequently used in cases of RDS, transient tachypnea of the newborn, pneumonia, and pneumothorax. Lung ultrasound has high specificity, sensitivity, positive predictive value, and negative predictive value. It is performed quickly at the bedside, allowing for rapid diagnosis and timely intervention.

Respiratory distress syndrome is one of the most common causes of morbidity and mortality in preterm infants. It results from a surfactant deficiency in the lungs secondary to preterm birth. Early diagnosis and timely administration of intratracheal surfactant, which is the only definitive treatment, are crucial. The diagnosis has traditionally relied on chest X-rays, but with recent advancements, lung ultrasound has also become a diagnostic tool. In addition to diagnosing RDS, lung ultrasound plays a critical role in its differential diagnosis, severity classification, and management in neonates.

Different methods can be used for the intratracheal administration of surfactant in the treatment of neonatal respiratory distress syndrome. Surfactant can be administered through an endotracheal tube in intubated infants. In non-intubated infants, two commonly accepted and frequently used methods are available. The first method involves intubating the infant, administering intratracheal surfactant, and then extubating them back to nasal respiratory support (ENSURE method). The second method involves delivering surfactant via a thin catheter (5F) directly into the trachea while the infant remains on existing nasal respiratory support, without disconnecting them from it (LISA method). Both of these methods are frequently used in neonatal intensive care units, and multiple studies comparing them indicate no clear superiority of one over the other.

Many studies utilizing lung ultrasound incorporate lung ultrasound scoring systems. The first neonatal lung ultrasound score was defined by Brat et al. Each lung is divided into three regions (upper anterior, lower anterior, and lateral), and each region is assigned a score from 0 to 3:

0 points: Defined by the presence of only A-lines.

1. point: Defined by the presence of three or more well-spaced B-lines.
2. points: Defined by the presence of multiple coalescing B-lines, with or without small subpleural consolidations.
3. points: Defined by the presence of large consolidation areas. The total score, obtained by summing the scores from all lung regions, represents the infant's overall lung ultrasound score. Scores range from 0 (completely normal) to 18.

Based on existing lung ultrasound studies, this study will evaluate preterm infants born before 32 weeks gestation who are diagnosed with RDS. Serial lung ultrasounds will be performed at different time points following surfactant administration (5 minutes, 10 minutes, 20 minutes, 30 minutes, 1 hour, 2 hours, and 6 hours after completion of surfactant administration), and lung ultrasound scores will be calculated. The aim is to determine whether different surfactant administration methods result in different lung ultrasound scores over time.

This study aims to investigate the relationship between the method of surfactant administration and improvements in serial lung ultrasound findings in preterm infants requiring surfactant therapy.

The investigators plan to conduct their study at Konya City Hospital between July 2024 and July 2025. Preterm infants born at their hospital at or below 32 weeks of gestation, diagnosed with RDS, and requiring surfactant therapy without intubation will be included in the study. The families of the infants planned for inclusion will be informed about the study, and written consent will be obtained if they agree to participate. Only infants whose families provide consent will be included. The follow-up process and treatments of the included infants will not be altered in any way. The method of surfactant administration will be determined by the attending neonatologist. The physician performing the ultrasound evaluations and the principal investigator will be blinded to the method of surfactant administration. The choice of surfactant administration method will be made solely by the responsible physician.

A total of seven serial lung ultrasound evaluations will be performed at 5 minutes, 10 minutes, 20 minutes, 30 minutes, 1 hour, 2 hours, and 6 hours after the completion of surfactant administration. Lung ultrasound scoring will be applied (each lung is divided into three regions: upper anterior, lower anterior, and lateral. Each region is assigned a score from 0 to 3: 0 points indicate the presence of only A-lines; 1 point indicates the presence of ≥3 well-spaced B-lines; 2 points indicate multiple coalescent B-lines, with or without subpleural consolidations; and 3 points indicate large consolidation areas). All ultrasound evaluations throughout the study will be performed by the same physician.

The demographic and clinical characteristics of the patients, as well as prenatal/postnatal risk factors, will be recorded in the patient data collection form. Additionally, ultrasound scoring results, oxygen requirements, and saturation values will be documented.

No invasive procedures will be performed on the patients, and no blood samples will be collected for the study.

ELIGIBILITY:
Inclusion Criteria:

* Infants of families who agree to participate in the study
* Preterm infants born before 32 weeks of gestation requiring surfactant therapy due to an RDS diagnosis.

Exclusion Criteria:

* Infants whose families did not provide consent
* Infants with a syndromic appearance or congenital heart disease
* Preterm infants born after 32 weeks of gestation

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 68 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of serial lung ultrasound data after surfactant treatments | 6 hours after completion of surfactant administration
  This study aims to investigate the relationship between the method of surfactant administration and improvements in serial lung ultrasound findings in preterm infants requiring surfactant therapy.

CONTACTS AND LOCATIONS:
Overall Officials: MELEK BUYUKEREN, Principal Investigator — Konya City Hospital
Locations (1):
- Melek Buyukeren, Konya, karatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Once the study is published as a scientific article, it can be shared.

REFERENCES:
- [Background] Avni EF, Braude P, Pardou A, Matos C. Hyaline membrane disease in the newborn: diagnosis by ultrasound. Pediatr Radiol. 1990;20(3):143-6. doi: 10.1007/BF02012957. PMID 2191263
- [Background] Corsini I, Parri N, Gozzini E, Coviello C, Leonardi V, Poggi C, Giacalone M, Bianconi T, Tofani L, Raimondi F, Dani C. Lung Ultrasound for the Differential Diagnosis of Respiratory Distress in Neonates. Neonatology. 2019;115(1):77-84. doi: 10.1159/000493001. Epub 2018 Oct 10. PMID 30304736
- [Background] Liu X, Si S, Guo Y, Wu H. Limitations of Bedside Lung Ultrasound in Neonatal Lung Diseases. Front Pediatr. 2022 Apr 26;10:855958. doi: 10.3389/fped.2022.855958. eCollection 2022. PMID 35558371
- [Background] Singh Y, Tissot C, Fraga MV, Yousef N, Cortes RG, Lopez J, Sanchez-de-Toledo J, Brierley J, Colunga JM, Raffaj D, Da Cruz E, Durand P, Kenderessy P, Lang HJ, Nishisaki A, Kneyber MC, Tissieres P, Conlon TW, De Luca D. International evidence-based guidelines on Point of Care Ultrasound (POCUS) for critically ill neonates and children issued by the POCUS Working Group of the European Society of Paediatric and Neonatal Intensive Care (ESPNIC). Crit Care. 2020 Feb 24;24(1):65. doi: 10.1186/s13054-020-2787-9. PMID 32093763
- [Background] Guo BB, Pang L, Yang B, Zhang C, Chen XY, OuYang JB, Wu CJ. Lung Ultrasound for the Diagnosis and Management of Neonatal Respiratory Distress Syndrome: A Minireview. Front Pediatr. 2022 Apr 14;10:864911. doi: 10.3389/fped.2022.864911. eCollection 2022. PMID 35498779
- [Background] Fortas F, Loi B, Centorrino R, Regiroli G, Ben-Ammar R, Shankar-Aguilera S, Yousef N, De Luca D. Enhanced INSURE (ENSURE): an updated and standardised reference for surfactant administration. Eur J Pediatr. 2022 Mar;181(3):1269-1275. doi: 10.1007/s00431-021-04301-x. Epub 2021 Nov 4. PMID 34735625
- [Background] Brat R, Yousef N, Klifa R, Reynaud S, Shankar Aguilera S, De Luca D. Lung Ultrasonography Score to Evaluate Oxygenation and Surfactant Need in Neonates Treated With Continuous Positive Airway Pressure. JAMA Pediatr. 2015 Aug;169(8):e151797. doi: 10.1001/jamapediatrics.2015.1797. Epub 2015 Aug 3. PMID 26237465
- [Background] Pareek P, Deshpande S, Suryawanshi P, Sah LK, Chetan C, Maheshwari R, More K. Less Invasive Surfactant Administration (LISA) vs. Intubation Surfactant Extubation (InSurE) in Preterm Infants with Respiratory Distress Syndrome: A Pilot Randomized Controlled Trial. J Trop Pediatr. 2021 Aug 27;67(4):fmab086. doi: 10.1093/tropej/fmab086. PMID 34595526